CLINICAL TRIAL: NCT01806766
Title: Comparison of Ceramic-on-Ceramic and Ceramic-on-Highly-Cross-Linked Polyethylene Bearings in Primary Cementless Total Hip Arthroplasty in the Same Patients
Brief Title: Comparison of Ceramic-on-Ceramic and Ceramic-on-Highly-Cross-Linked Polyethylene Bearings
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ewha Womans University (Other)
Responsible Party: Principal Investigator, Young Hoo Kim, Professor, Ewha Womans University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XPECCC
Record Dates: First submitted 2013-03-05; First posted 2013-03-07 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Osteonecrosis; Osteoarthritis
Keywords: cementless total hip arthroplasty; ceramic on ceramic bearing; ceramic on highly cross linked polyethylene; young patient
MeSH Terms: conditions — Osteonecrosis; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ceramic on Ceramic (Active Comparator): Ceramic on Ceramic bearing coupled side of a single patient undergoing bilateral total hip arthroplasty
  Interventions: Procedure: Ceramic on Ceramic bearing
- Ceramic on HXPE (Active Comparator): Ceramic on HIghly crosslinked polyethylene bearing coupled side of a single patient undergoing bilateral total hip arthroplasty
  Interventions: Procedure: Ceramic on Highly crosslinked polyethylene bearing

INTERVENTIONS:
Procedure: Ceramic on Ceramic bearing — cementless Total Hip Arthroplasty with Ceramic on ceramic bearing
  Arms: Ceramic on Ceramic
Procedure: Ceramic on Highly crosslinked polyethylene bearing — Cementless Total Hip Arthroplasty with Ceramic on Highly crosslinked polyethylene bearing
  Arms: Ceramic on HXPE

SUMMARY:
The purpose of this prospective, randomized study was to compare the clinical and radiographic results and the prevalence of osteolysis of the cementless total hip arthroplasty with an alumina-on-alumina bearings one side and alumina-on-highly cross-linked polyethylene bearings on the other side in the young and active patients.

ELIGIBILITY:
Inclusion Criteria:

* Primary hip osteoarthritis
* Secondary hip osteoarthritis
* Avascular necrosis of femoral head

Exclusion Criteria:

* Previous surgical history of hip

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 1998-01; Primary Completion 2000-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Harris hip score | Pre-op, last follow-up(11-13 years)
  Comparing harris hip score before and after the intervention, and at the final follow-up, between two sides.

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index(WOMAC) | preop, last follow-up(11-13 years)
  WOMAC index before, and after the intervention, and between sides at the last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Young-Hoo Kim, MD, Study Director — Ewha Womans University Mokdong Hospital
Locations (1):
- Ewha Womans University Mokdong Hospital, Seoul, South Korea